CLINICAL TRIAL: NCT03232424
Title: Pilot Study of Concomitant NovoTTF-200A and Temozolomide Chemoradiation for Newly Diagnosed Glioblastoma
Brief Title: NovoTTF-200A and Temozolomide Chemoradiation for Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2017-0087
Record Dates: First submitted 2017-07-17; First posted 2017-07-28 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Glioblastoma, Adult
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: Prospective, single arm, non-randomized, open label pilot
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- NovoTTF-200A + Temozolomide Chemoradiation (Experimental): NovoTTF-200A, concomitant with radiotherapy and temozolomide, as front-line therapy for glioblastoma
  Interventions: Device: NovoTTF-200A; Drug: Temozolomide; Radiation: 3D conformal or intensity modulated radiation therapy (IMRT)

INTERVENTIONS:
Device: NovoTTF-200A — * Begins the day prior to radiotherapy start and continues until the end of temozolomide maintenance cycle #2 or until evidence of disease progression or unacceptable toxicity.
  * Arrays are removed immediately prior to radiotherapy and replaced immediately thereafter.
  Other Names: Optune
Drug: Temozolomide — Concomitant phase:
  * 75 mg/m2 per day for 42 days concomitant with radiotherapy.
  * Begins 1 day prior to XRT start.
  Maintenance phase:
  * Begins 4 weeks after concomitant phase completion (+/- 1 week).
  * Each cycle is 28 days (5 days of drug treatment followed by 23 days without).
  * Cycle 1: 150 mg/m2 once daily for the first 5 days of each treatment cycle.
  * Subsequent cycles: daily dose increased to 200 mg/m2, if the CTC non-hematologic toxicity for Cycle 1 is Grade ≤ 2 (except for alopecia, nausea and vomiting), absolute neutrophil count (ANC) is ≥ 1.5 x 109/L, and the platelet count is ≥ 100 x 109/L. The dose remains at 200 mg/m2 per day for the first 5 days of each subsequent cycle except if toxicity occurs.
Radiation: 3D conformal or intensity modulated radiation therapy (IMRT) — Radiotherapy will commence 4 weeks after the definitive surgical procedure (+/- 1 week), to a total dose of 54.0 - 60.0 Gy, delivered in 1.8 - 2.0 Gy fractions over 6 - 7 weeks. XRT target volumes will be determined utilizing all available imaging studies that best delineate extent of disease. Fusion image registration for treatment planning will be utilized as possible. Either 3D conformal or intensity modulated radiation therapy (IMRT) will be utilized.

SUMMARY:
This study is a prospective single arm trial designed to study the safety, feasibility and preliminary efficacy of a medical device, NovoTTF-200A used concomitantly with standard adjuvant treatment for newly diagnosed glioblastoma.

DETAILED DESCRIPTION:
A prospective, single arm, non-randomized, open label pilot trial will enroll ten patients with histologically-confirmed newly diagnosed GBM who meet all eligibility criteria. Patients will be recruited to the study by the principal investigator (PI) or one of the co-investigators (CI) at one institution, Hackensack University Medical Center. Accrual is expected to continue for 18 months.

The protocol has a planned enrollment of 10 patients. Should patients discontinue treatment on protocol for reasons unrelated to toxicity (e.g. lost to follow-up, withdrawal of consent), additional patient (s) may be enrolled to complete enrollment.

Following maximal debulking surgery, patients will undergo a gadolinium enhanced brain MRI within 72 hours and a screening visit 2 to 4 weeks following surgery. Extent of resection will be recorded as biopsy, partial resection or gross-total resection based upon residual enhancing tumor on post-operative MRI.The day prior to XRT start, patients will have a clinic visit for training and application of the NovoTTF-200A device. During this visit, the patient will be educated regarding general use and maintenance of the device, with a particular focus upon strategies to prevent, identify and manage dermatologic adverse events (dAE). Temozolomide will be dosed nightly during XRT as per standard of care, and NovoTTF-200A will be worn continuously, removed during XRT and replaced as soon as possible thereafter.

During XRT and for 12 weeks to follow, the patient will have study visits at regular intervals (TAB A) for a physical examination and to assess toxicity and device compliance. Visits outlined in TAB A are in addition to weekly visits during radiotherapy with the treating radiation oncologist. MRI will be obtained at 4 weeks (+/-7 days) and 12 weeks (+/-7 days) following completion of XRT, and maintenance temozolomide will recommence in 5/28 day cycles as per standard of care. Objective response will be assessed as defined by the Response Assessment in Neuro-Oncology (RANO) criteria (TAB C) by the treating physician and confirmed by a second investigator.

In the case of suspected pseudoprogression, continued treatment and subsequent evaluations will help clarify whether it is true progression. Patients may continue treatment at the discretion of the investigator. If subsequent evaluations suggest that the tumor has in fact progressed, the date of progression will reflex to the date when the issue was first raised. However, if subsequent evaluations demonstrate improvement without change in therapy, the initial tumor increase may be considered pseudoprogression and response may be recorded as not evaluable for that time point. In the case of clinical progression, an unscheduled MRI will be obtained within 1 week of the investigator becoming aware of the clinical progression. No additional MRIs will be required after progression.

Temozolomide and NovoTTF-200A will continue until the final study visit, or until disease progression or unacceptable toxicity. Thereafter, temozolomide, MRI and response assessments will continue as per standard of care. Following the final study visit, the patient will be followed at a minimum of every two months for survival, either by phone or in person. If the patient is free of unacceptable toxicity attributable to NovoTTF-200A, they will be offered the opportunity to continue the device at no financial cost, but without obligation to do so.

Unacceptable toxicity includes the occurrence of device related serious adverse events or clinical and functional deterioration considered by the investigator to be prohibitive of continuing treatment. Treatment with the NovoTTF-200A device does not need to be terminated in the case of temozolomide toxicity.

The primary endpoint will be safety and tolerability of combined modality treatment with radiotherapy, temozolomide and NovoTTF-200A, based upon the incidence and severity of adverse events. Secondary endpoints will be overall survival, progression free survival and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed GBM using WHO criteria.
2. Age ≥ 18 years
3. Maximal debulking surgery (at the discretion of the investigator). Biopsy alone is not exclusionary.
4. KPS ≥ 70
5. Life expectancy of at least 3 months.
6. Sexually active participants must agree to the strict use of barrier contraception.
7. Patients must be able to understand the investigational nature of the study and provide informed consent.
8. Adequate hematologic function:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   2. Platelet count ) ≥ 100 x 109/L
   3. Hemoglobin ≥ 10 g /dL
9. Adequate liver function

   1. Total bilirubin ≤ 1.5 x ULN
   2. AST and ALT ≤ 2.5 x ULN
10. Adequate renal function

    a. Creatinine ≤ 1.25 x ULN
11. International normalized ratio (INR) or PT and activated partial thromboplastin time (aPTT): 1.5 x ULN (except for subjects receiving anticoagulation therapy). Use of anticoagulants is permitted as long as the INR or aPTT are within therapeutic limits (according to the medical standard of the institution).

Exclusion Criteria:

1. Active participation in another clinical treatment trial. Concomitant protocols for data or tissue collection without intervention are permitted.
2. Any prior treatment for GBM aside from surgery, including carmustine wafers.
3. Women who are pregnant or nursing.
4. Severe acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with trial participation, NovoTTF-200A device use or interfere with interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into the trial. This includes but not limited to:

   1. Patients with inadequately healed surgical incisions or other dermatologic scalp toxicity at baseline (grade 2 or higher, as defined in Section VIII) upon which transducer leads may require placement.
   2. Known HIV or other immunosuppressive disease, chronic hepatitis B or hepatitis C
   3. Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of the protocol.
5. Implanted pacemaker, programmable shunt, cardiac defibrillator, deep brain stimulator, other implanted electronic devices in the brain or documented clinically significant arrhythmias.
6. Infratentorial glioblastoma.
7. Past hypersensitivity reaction to temozolomide or DTIC.
8. Psychiatric illness that compromises the informed consent process, at the discretion of the investigator.
9. Inability or unwillingness to return for required visits.
10. Previous cytotoxic therapy within the last 5 years.
11. Inability to begin temozolomide concomitant to radiation therapy, for reasons 4 or 7 above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 24 months
  Safety and tolerability of combined modality treatment with radiotherapy, temozolomide and NovoTTF-200A based upon the incidence and severity of adverse events.

SECONDARY OUTCOMES:
Overall survival time | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  Assessed from NovoTTF-200A start date to date of death of any cause. Patients will be censored at the time that they are last known to be alive (if withdrawn or lost to follow-up).
Progression free survival at 6 months | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  Assessed from NovoTTF-200A start date to the date of the first observation of clinical or radiographic disease progression or death due to any cause. Patients will be censored at the time they are last known to be alive and progression free (if withdrawn or lost to follow-up).
Quality of life assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of life questionnaire (QLQ-C30) | 24 months
  Change from baseline at each measure will be calculated for each subscale domain and symptom scale in the questionnaire. The QLQ-C30 incorporates five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status / QoL scale, and a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnea, loss of appetite, insomnia, constipation and diarrhea) and perceived financial impact of the disease. The response scale to each question ranges from 1 (Not at All) to 4 (Very Much). For each subscale domain and symptom scale, the change from baseline will summarized as mean (SD) or median (interquartile range), as appropriate.
Quality of life assessed using a European Organization for Research and Treatment of Cancer (EORTC) Brain Cancer questionnaire (BN20) | 24 months
  Change from baseline at each measure will be calculated for each subscale domain and symptom scale in the questionnaire. The questionnaire includes 20 items assessing future uncertainty, visual disorder, motor dysfunction, communication deficit and other disease symptoms (e.g. headaches and seizures) and treatment toxicities (e.g. hair loss). The response scale to each question ranges from 1 (Not at All) to 4 (Very Much). For each subscale domain and symptom scale, the change from baseline will summarized as mean (SD) or median (interquartile range), as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Goldlust, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895
- [Background] Polk C. Therapeutic applications of low-frequency sinusoidal and pulsed electric and magnetic fields. In: Bronzino JD ed. The biomedical engineering handbook. Connecticut: CRC Press, 1995:1404-1416.
- [Background] Palti Y. Stimulation of internal organs by means of externally applied electrodes. J Appl Physiol. 1966 Sep;21(5):1619-23. doi: 10.1152/jappl.1966.21.5.1619. No abstract available. PMID 5923236
- [Background] Bassett CA. The development and application of pulsed electromagnetic fields (PEMFs) for ununited fractures and arthrodeses. Clin Plast Surg. 1985 Apr;12(2):259-77. PMID 3886262
- [Background] Elson E. Biologic Effects of radiofrequency and microwave fields: in vivo and in vitro experimental results. In: Bronzino JD ed. The biomedical engineering handbook. Connecticut: CRC Press, 1995:1417-1423.
- [Background] Chou CK. Radiofrequency hyperthermia in cancer therapy. In: Bronzino JD ed. The biomedical engineering handbook. Connecticut: CRC Press, 1995:1424-1430.
- [Background] Takashima S, Schwan HP. Alignment of microscopic particles in electric fields and its biological implications. Biophys J. 1985 Apr;47(4):513-8. doi: 10.1016/S0006-3495(85)83945-X. PMID 3986280
- [Background] Zimmermann U, Vienken J, Pilwat G. Rotation of cells in an alternating electric field: the occurrence of a resonance frequency. Z Naturforsch C Biosci. 1981 Jan-Feb;36(1-2):173-7. doi: 10.1515/znc-1981-1-229. PMID 7010816
- [Background] Holzapfel C, Vienken J, Zimmermann U. Rotation of cells in an alternating electric field: theory and experimental proof. J Membr Biol. 1982;67(1):13-26. doi: 10.1007/BF01868644. PMID 7097755
- [Background] Pawlowski P, Szutowicz I, Marszalek P, Fikus M. Bioelectrorheological model of the cell. 5. Electrodestruction of cellular membrane in alternating electric field. Biophys J. 1993 Jul;65(1):541-9. doi: 10.1016/S0006-3495(93)81056-7. PMID 8369458
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Zhao M, Forrester JV, McCaig CD. A small, physiological electric field orients cell division. Proc Natl Acad Sci U S A. 1999 Apr 27;96(9):4942-6. doi: 10.1073/pnas.96.9.4942. PMID 10220398
- [Background] Jordan MA, Thrower D, Wilson L. Effects of vinblastine, podophyllotoxin and nocodazole on mitotic spindles. Implications for the role of microtubule dynamics in mitosis. J Cell Sci. 1992 Jul;102 ( Pt 3):401-16. doi: 10.1242/jcs.102.3.401. PMID 1506423
- [Background] Rowinsky EK, Donehower RC. Paclitaxel (taxol). N Engl J Med. 1995 Apr 13;332(15):1004-14. doi: 10.1056/NEJM199504133321507. No abstract available. PMID 7885406
- [Background] Kline-Smith SL, Walczak CE. The microtubule-destabilizing kinesin XKCM1 regulates microtubule dynamic instability in cells. Mol Biol Cell. 2002 Aug;13(8):2718-31. doi: 10.1091/mbc.e01-12-0143. PMID 12181341
- [Background] Kapoor TM, Mayer TU, Coughlin ML, Mitchison TJ. Probing spindle assembly mechanisms with monastrol, a small molecule inhibitor of the mitotic kinesin, Eg5. J Cell Biol. 2000 Sep 4;150(5):975-88. doi: 10.1083/jcb.150.5.975. PMID 10973989
- [Background] Maiato H, Sampaio P, Lemos CL, Findlay J, Carmena M, Earnshaw WC, Sunkel CE. MAST/Orbit has a role in microtubule-kinetochore attachment and is essential for chromosome alignment and maintenance of spindle bipolarity. J Cell Biol. 2002 May 27;157(5):749-60. doi: 10.1083/jcb.200201101. Epub 2002 May 28. PMID 12034769
- [Background] Gagliardi LJ. Electrostatic force in prometaphase, metaphase, and anaphase-A chromosome motions. Phys Rev E Stat Nonlin Soft Matter Phys. 2002 Jul;66(1 Pt 1):011901. doi: 10.1103/PhysRevE.66.011901. Epub 2002 Jul 12. PMID 12241378
- [Background] Fishkind DJ, Silverman JD, Wang YL. Function of spindle microtubules in directing cortical movement and actin filament organization in dividing cultured cells. J Cell Sci. 1996 Aug;109 ( Pt 8):2041-51. doi: 10.1242/jcs.109.8.2041. PMID 8856500
- [Background] Dogterom M, Yurke B. Measurement of the force-velocity relation for growing microtubules. Science. 1997 Oct 31;278(5339):856-60. doi: 10.1126/science.278.5339.856. PMID 9346483
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Kirson ED, Schneiderman RS, Dbaly V, Tovarys F, Vymazal J, Itzhaki A, Mordechovich D, Gurvich Z, Shmueli E, Goldsher D, Wasserman Y, Palti Y. Chemotherapeutic treatment efficacy and sensitivity are increased by adjuvant alternating electric fields (TTFields). BMC Med Phys. 2009 Jan 8;9:1. doi: 10.1186/1756-6649-9-1. PMID 19133110
- [Background] Stupp R, Wong E, Scott C et al. Interim analysis of the EF-14 trial: a prospective, multi-center trial of NovoTTF-100A together with temozolomide compared to temozolomide alone in patients with newly diagnosed GBM. Neuro Oncol 2014;16(suppl 5):v167.
- [Background] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262
- [Background] Pless M, Droege C, von Moos R, Salzberg M, Betticher D. A phase I/II trial of Tumor Treating Fields (TTFields) therapy in combination with pemetrexed for advanced non-small cell lung cancer. Lung Cancer. 2013 Sep;81(3):445-450. doi: 10.1016/j.lungcan.2013.06.025. Epub 2013 Jul 23. PMID 23891283
- [Background] Giladi M, Zielinska-Chomej K, Tichon A et al. The effect of alternating electric fields (TTFields) on inhibition of repair of DNA damage induced by ionizing radiation and sensitization of glioma and non-small cell lung cancer cells to radiation. J Clin Oncol 2014;32(suppl;abstr e22239).
- [Background] Zielinska-Chomej K, Grozman V, Tu J, Viktorsson K, Lewensohn R. Analysis of combination of tumor treating fields (TTFields) with radiotherapy in non-small cell lung cancer. Neuro Oncol 2013;15(suppl 3):ET-033.
- [Background] Lacouture ME, Davis ME, Elzinga G, Butowski N, Tran D, Villano JL, DiMeglio L, Davies AM, Wong ET. Characterization and management of dermatologic adverse events with the NovoTTF-100A System, a novel anti-mitotic electric field device for the treatment of recurrent glioblastoma. Semin Oncol. 2014 Jun;41 Suppl 4:S1-14. doi: 10.1053/j.seminoncol.2014.03.011. Epub 2014 Mar 19. PMID 24794308